CLINICAL TRIAL: NCT01357018
Title: A Study on Quality of Life in Patients With Chronic Arthritis
Brief Title: Quality of Life in Chronic Arthritis
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Sheng Wu, Chief, Division of Rheumatology, Far Eastern Memorial Hospital
Other Study IDs: 099094-E
Record Dates: First submitted 2010-12-07; First posted 2011-05-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Ankylosing Spondylitis; Rheumatoid Arthritis
Keywords: Ankylosing spondylitis; Disease activity; EQ-5D; Quality of life; Rheumatoid arthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with rheumatoid arthritis
- patients with ankylosing spondylitis

SUMMARY:
Chronic joint complaints are prevalent in clinical practice. If chronic arthritis such as rheumatoid arthritis (RA) or ankylosing spondylitis (AS) is not adequately controlled, it can not only affect patient's working ability but also produce indirect cost in patient's family. Quality of life will also be affected. Health-related quality of life issues are assuming increasing importance in chronic rheumatic diseases. However, studies on quality of life in rheumatic patients are limited. Factors related to quality of life are not clear. Application of quality of life measurement for improving clinical care of RA and AS patients is still difficult. The objective of this study was to evaluation the validity of EQ-5D life quality measurement in chronic arthritis patients in Taiwan. Factors associated with life quality will be addressed. This will also provide useful information for public health policy making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis or ankylosing spondylitis

Exclusion Criteria:

* Patients with mental illness which interfered with questionaire answering

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with rheumatoid arthritis or ankylosing spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Validity of life quality measurement EQ-5D in chronic arthritis patients | EQ-5D at recruitment and 6 months later in chronic arthritis patients
  Effect of age, gender, diagnosis, disease duration and education on subjective feeling of quality of life (by EQ-5D) will be analyzed. Repeated measurements will be used for analysis of association between disease activity and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Sheng Wu, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Taiwan